CLINICAL TRIAL: NCT02900950
Title: Multicolour Versus Monocolour Inking Specimens After Pancreaticoduodenectomy for Periampullary Cancer: a Single Center Prospective Randomised Clinical Trial.
Brief Title: Multicolour Versus Monocolour Specimens Inking After Pancreaticoduodenectomy for Periampullary Cancer
Acronym: MPM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Riccardo Casadei, Associate Professor of Surgery at University of Bologna, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: MPM-DCP
Record Dates: First submitted 2016-09-01; First posted 2016-09-15 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-09

CONDITIONS: Stage, Pancreatic Cancer; Neoplasm, Residual; Pancreatic Neoplasm; Periampullary Cancer
Keywords: cancer; resection margin; pathology; pancreas
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasm, Residual; Neoplasms; Margins of Excision

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A-Multicolour inking specimen (Experimental): After performing the pancreaticoduodenectomies, the surgeon intraoperatively inked the surfaces/margins of the specimen with different colours. The surfaces/margins inked were the following:
  1. Anterior surface of the pancreas (yellow);
  2. Posterior surface of the pancreas (orange);
  3. Superior mesenteric/portal vein groove (blu);
  4. Superior mesenteric artery margin (retroperitoneal margin) (red);
  5. Transection margin of the bile duct (green) The trans-section pancreatic and gastric margins were not inked.
  Interventions: Procedure: Multicolour inking specimens
- Arm B-Monocolour inking specimen (Other): In arm B, only the superior mesenteric artery margin and the pancreatic margin were intraoperatively indicated by the surgeon in the specimen: a single stitch to identify the transection pancreatic margin and a continuous suture to identify the superior mesenteric artery margin. Monochromatic inking of the superior mesenteric artery margin was subsequently carried out by the pathologist.
  Interventions: Procedure: Monocolour inking specimens

INTERVENTIONS:
Procedure: Multicolour inking specimens
  Arms: Arm A-Multicolour inking specimen
Procedure: Monocolour inking specimens
  Arms: Arm B-Monocolour inking specimen

SUMMARY:
A single-centre, randomised clinical trial of patients affected by periampullary cancer who underwent pancreaticoduodenectomies which included two different types of specimen margination: arm A (multicolour inking) and arm B (monocolour inking). The randomisation of the specimen was made after the resection, blinded for the surgeons involved in the operation. The primary endpoint was the overall R1 resection rate and its difference between the two arms. The secondary endpoints were the R1 resection rate in each margin and its difference between the two arms, and the impact of margin status on survival. A sample size of 18 patients was required.

DETAILED DESCRIPTION:
This study was a single-centre, prospective, controlled, open, parallel group, randomised clinical trial, conducted in the tertiary referral University Centre of S.Orsola-Malpighi Hospital, Bologna, Italy, from June 2012 to January 2016, which enrolled patients affected by periampullary cancer who underwent pancreaticoduodenectomy (PD). All patients with suspected periampullary cancer were enrolled in the study, but only patients who underwent pancreaticoduodenectomy were randomised and allocated to a multicolour inking specimen (arm A, experimental) or a monocolour inking (arm B, control) after specimen was taken out from the operative field. The analysis regarded only the specimens of the patients who underwent PD in which the final pathologic report showed a diagnosis of invasive periampullary cancer (pancreatic, ampullary and distal bile duct).

After performing the pancreaticoduodenectomies, the surgeon intraoperatively inked the surfaces/margins of the specimen with different colours. In the multicolour arm, the surfaces/margins inked were the following: Anterior surface of the pancreas (yellow); Posterior surface of the pancreas (orange); Superior mesenteric/portal vein groove (blu); Superior mesenteric artery margin (retroperitoneal margin) (red); Transection margin of the bile duct (green).The trans-section pancreatic and gastric margins were not inked.

In the monocolour arm, only the superior mesenteric artery margin and the pancreatic margin were intraoperatively indicated by the surgeon in the specimen: a single stitch to identify the transection pancreatic margin and a continuous suture to identify the superior mesenteric artery margin. Monochromatic inking of the superior mesenteric artery margin was subsequently carried out by the pathologist. In both arms of treatment, the macroscopic evaluation and slicing of the surgical specimen followed the Leeds Pathology Protocol (LEEPP), and seven margins, which included the anterior, posterior, superior mesenteric /portal vein groove, superior mesenteric artery, bile duct, pancreatic neck and stomach margins, were examined. The primary endpoint was to evaluate the overall R1 resection rate and its difference between multicolour (arm A) and monocolour (arm B) inking of the specimen. The secondary endpoints were to evaluate the R1 resection rate in each margin: anterior and posterior surfaces of the pancreatic head; superior mesenteric/portal vein groove; superior mesenteric artery margin; transection pancreatic and bile duct margins, and its difference between the two arms compared. Finally, the impact of the margin status on survival was considered for each margin and type of periampullary tumours.

Calculation of the sample size was based on the literature assumption that the overall incidence rate expected of R1 ranged from 10 to 76% while it increased to 81-85% when a standardised pathological technique and margination with multicolour inking, as described in arm A, was performed. To detect a difference in R1 rate between these values with a 5% alpha-error and a 80% beta-error at a two-sided 0.05 significance level, a sample size of 18 patients was required for each group. In relation to the fact that the patients were often randomised without a preoperative biopsy, and that following current literature the 5-13% of the presumed malignancies were benign, it was decided to randomise 25 patients in order to avoid a sample size smaller than expected. The sample size calculation was carried out using PS Power and Sample Size Calculation software (Department of Biostatistics; Vanderbilt University; Nashville, TN, USA).

ELIGIBILITY:
Inclusion Criteria:

* medical history without previous pancreatic resection or pancreatic cancer
* written consent

Exclusion Criteria:

* patients previously treated with chemotherapy radiotherapy or chemoradiotherapy for pancreatic cancer
* patients with diagnostic doubts of chronic pancreatitis, serous cystic tumours, intraductal papillary mucinous tumours or neuroendocrine tumours
* patients unresectable at laparotomy
* patients who had undergone other pancreatic resections (total or subtotal pancreatectomy).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2012-06; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Evaluate overall microscopic resection margins involvement (R1 rate) after pancreaticoduodenectomy for periampullary cancer. | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.
Evaluate R1 rate differences between multicolour and monocolour inking of the specimen | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.

SECONDARY OUTCOMES:
Evaluate R1 resection rate in anterior surface of the pancreatic head. | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.
Evaluate R1 resection rate in posterior surface of the pancreatic head. | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.
Evaluate R1 resection rate in superior mesenteric/portal vein groove | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.
Evaluate R1 resection rate in superior mesenteric artery margin | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.
Evaluate R1 resection rate in pancreatic transection margin | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.
Evaluate R1 resection rate in common bile duct margin | At the time of pathological examination
  Microscopic margin involvement (R1) was defined as a distance of the tumour from the resection margin of ≤1 mm.
Disease Free Survival and Overall Survival of the participants | Through study completion, an average of 6 months
  Disease Free Survival and Overall Survival of the participants are measured using Kaplan-Meier curves.
Relation between Disease Free Survival and Overall Survival of the participants and R status | Through study completion, an average of 6 months
  Disease Free Survival and Overall Survival of the participants are measured using Kaplan-Meier curves and divided in subgroups related to their margin status (R0 versus R1).

CONTACTS AND LOCATIONS:
Overall Officials: Riccardo Casadei, Professor, Principal Investigator — S. Orsola-Malpighi Hospita, University of Bologna, Italy
Locations (1):
- S.Orsola-Malpighi Hospital, University of Bologna, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No